CLINICAL TRIAL: NCT05362032
Title: Feasibility of OmnEcoil System for Integrated Endorectal MRI and Transrectal MRI-Targeted Biopsy of the Prostate
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team paused enrollment
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Fergus Coakley, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00019964; NCI-2021-03941 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00019964 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2022-04-21; First posted 2022-05-05 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (endorectal MRI, MRI-targeted biopsy) (Experimental): Patients undergo endorectal MRI and transrectal MRI-targeted biopsy using the OmnEcoil device.
  Interventions: Device: Biopsy; Procedure: Endorectal Magnetic Resonance Imaging

INTERVENTIONS:
Device: Biopsy — Undergo transrectal MRI-targeted biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Endorectal Magnetic Resonance Imaging — Endorectal MRI
  Other Names: Endorectal MRI

SUMMARY:
This clinical trial tests whether it is feasible to use the OmnEcoil system for transrectal magnetic resonance imaging (MRI) to visualize and biopsy suspicious lesions in the prostate. The OmnEcoil device combines an endorectal coil (a type of wire placed within the rectum during diagnostic endorectal MRI to take better images of the prostate) with an endorectal probe. The OmnEcoil system is designed to allow for MRI to be used at the same time to image the prostate and aid in the biopsy of the suspected prostate cancer. Usually, these are performed as two separate events at two separate times.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate that the OmnEcoil system can obtain diagnostic tissue samples in vivo. (Early Feasibility Study)

II. To evaluate physician experience using OmnEcoil system. (Early Feasibility Study)

III. To monitor the safety of the OmnEcoil system. (Early Feasibility Study)

IV. To determine the performance of the OmnEcoil system as measured by the acquisition of diagnostic tissue samples and cancer containing biopsies of target lesions. (Traditional Feasibility Study)

V. To monitor the safety of the OmnEcoil system. (Traditional Feasibility Study)

EXPLORATORY OBJECTIVES:

I. To evaluate participant comfort after undergoing MRI-targeted prostate biopsy using OmnEcoil. (Early and Traditional Feasibility)

II. To assess the time required in the MRI scanner to perform an integrated MRI and biopsy using the OmnEcoil system. (Early and Traditional Feasibility)

OUTLINE:

Patients undergo endorectal MRI and transrectal MRI-targeted biopsy using the OmnEcoil device.

ELIGIBILITY:
Inclusion Criteria:

* Males, aged >= 45 years
* Willing and able to provide written informed consent, including willingness to undergo MRI-targeted biopsy using OmnEcoil investigational system
* Persistently elevated (> 3 ng/mL) or rising prostate specific antigen (PSA) level and/or abnormal digital rectal exam
* Prior negative transrectal ultrasound (TRUS) biopsy, or prior TRUS biopsy or transurethral resection of the prostate showing Gleason score =< 6 disease
* Received multiparametric prostate MRI within last 6 months prior to study enrollment with images available on Oregon Health and Science University (OHSU) image viewing system for review
* Must have at least one high-value biopsy target (i.e., score of 4 or 5 as categorized by Prostate Imaging and Reporting and Data System [PI-RADS] version 2.1) present on multiparametric MRI as evaluated by study radiologists
* Eastern Cooperative Group (ECOG) performance score 0 or 1
* Patient able to lie prone in MRI for OmnEcoil biopsy procedure
* Considered to be low bleeding risk [per Society for Interventional Radiology], including:

  * International normalized ratio (INR) <= 1.5, and
  * Platelets >= 50,000

Exclusion Criteria:

* Contraindication to MRI (e.g., severe claustrophobia, intracranial aneurysm clips, intraocular metallic foreign body, and cardiac pacemaker)
* Any contraindication to endorectal devices and/or biopsy, including (but not limited to) severe hemorrhoids, anal fissure, recent rectal surgery, or prior abdominoperineal resection
* Any bleeding diathesis and/or anti-coagulative therapy that cannot be temporarily reversed
* Active infection requiring systemic antibiotic therapy. Participants requiring systemic antibiotics for infection must have completed antibiotic therapy before initiating OmnEcoil imaging/biopsy procedure
* Administration of treatment for prostate cancer such as radiation or hormonal therapy prior to MRI-targeted biopsy
* Uncontrolled intercurrent illness that would substantially increase risk of incurring adverse events (AEs), confound results, or compromise the ability of the patient to give written informed consent
* Subjects unwilling to accept a blood transfusion

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Successful acquisition of tissue samples (early feasibility study) | Start of procedure to end of procedure, an average of less than 1 day
  Conducted with 10 subjects to demonstrate that OmnEcoil system can be used to obtain diagnostic tissue samples.
Physician device-user scores (early feasibility study) | Start of procedure to end of procedure, an average of less than 1 day
  Physician will rate device using a scale from 1 (excellent) to 5 (poor) following completion of OmnEcoil guided biopsy.
Incidence of biopsy-related grade >= 3 adverse events (early feasibility study) | Up to 30 days after end of procedure
  Assessed per Common Terminology Criteria for Adverse Events version 5.0.
Successful acquisition of diagnostic tissue samples (traditional feasibility study) | Start of procedure to end of procedure, an average of less than 1 day
  Procedure success determined by pathological review establishing that the samples are adequate for diagnosis. Criteria for acceptance is success rate >= 90%.
Presence of cancer containing biopsies of dominant targets (traditional feasibility study) | Start of procedure to end of procedure, an average of less than 1 day
  Criteria for acceptance is proportion of cancer containing biopsies >= 76%.
Incidence of biopsy-related grade >= 3 adverse events (traditional feasibility study) | Up to 30 days after end of procedure
  Assessed per Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Fergus V Coakley, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States